CLINICAL TRIAL: NCT04284969
Title: Prehabilitation & Rehabilitation in Oncogeriatrics: Adaptation to Deconditioning Risk and Accompaniment of Patients' Trajectories-ovary/Elderly Women With Ovarian Cancer-2, a GINECO Multicenter Randomized Study (PROADAPT-ovary/EWOC-2)
Brief Title: PROADAPT-ovary/EWOC-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL18_0359
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Surgery
Keywords: Cytoreductive surgery; Older; Senior adult; Prehabilitation
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients treated according current practice of the inclusion center. If interventions are implemented locally (geriatric assessment, nutrition, physical activity) they may be proposed to the patient.
- Intervention arm : PROADAPT program (Experimental): Patients benefiting from the PROADAPT (interventional arm) program.
  Interventions: Behavioral: PROADAPT program

INTERVENTIONS:
Behavioral: PROADAPT program — * A pre-intervention activity by telephone follow-ups every week for 12 weeks and then every month.
  * Pre-operative physical training including strength, endurance and breathing exercises.
  * A nutrition activity.
  * An activity to educate patients (on nutrition, exercise).
  * The implementation of standardised intervention procedures, established in agreement with the surgeons' representatives.
  * A pharmaceutical drug conciliation activity: optimization of the patient's different treatments with pharmaceutical expertise.
  * A transition activity from the hospital to the home, and a telephone follow-up up to 12 weeks after the surgery.
  Arms: Intervention arm : PROADAPT program

SUMMARY:
PROADAPT is a standardized geriatric intervention that is currently being co-constructed during an exploratory phase on a multi-professional and multi-disciplinary basis after a systematic analysis of published data (Figure).

It consists in: 1) before surgery: a prehabilitation of the patients including a nutritional, physical and educational preparation; 2) during the hospitalization for surgery: an optimisation of their treatments through a pharmaceutical conciliation, educational interventions, standardization of surgical procedures and enhanced rehabilitation after surgery; 3) bridging and post-discharge interventions for hospital-to-home transition.

This intervention is based on a logic change model, constructed with literature data and validated by an expert group through a DELPHI method : the rehabilitation model.

This intervention was designed to be implemented pragmatically in the centers according local habits and is currently being evaluated in several distinct hospital contexts under the name of "PROADAPT pilot study" in different tumor contexts thanks to a grant from the Regional Health Agency of Rhône-Alpes Auvergne region.

PROADAPT intervention is planned to be evaluated in 4 tumor models inducing complex medico-surgical procedures considered at high risk of geriatric deconditioning. They have the same primary objectives in order to be evaluated into a meta-analysis. Results will be used to test the validity of the rehabilitation model. Therefore, it is a study reaching the goal of the population health intervention research.

The purpose of the PROADAPT-ovary/EWOC-2 study is to evaluate the impact of PROADAPT on patient's post-surgical outcomes in patients ≥ 70 years old with an advanced ovarian cancer (AOC).

DETAILED DESCRIPTION:
With the conjunction of increased life expectancy and the increasing incidence of cancer with aging, older patient represent an increasing proportion of cancer patients. Increasing age is also associated with increased risk of co-morbidities as well as a decline of functional reserve of multiple organ systems, eventually leading in the context of the disease-and/or the treatment-related stress to functional deconditioning or organ failure.

Surgery or complex medico-surgical procedures can be considered as one proof-of principle of such risks, since major cancer surgery the older population is at higher risk of morbi-mortality and unplanned hospitalization for geriatric events1.

In order to reduce complications after surgery, prehabilitation has often been considered, and 71% of the surgeons would accept a 4 weeks delay before surgery to improve patients' outcomes if shown to be beneficial2. However, the actual level of evidence depends on the interventions: high for pre-operative nutrition3, but low for physical exercise, due to heterogeneous programs with often bad adherence4. In addition, geriatric validated interventions, in order to prevent iatrogenic event, may be added in a multi-interventional model of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥70 year old OR Woman ≥60 years with significant comorbid condition (modified Charlson index≥3) or disability (ADL score<6/6);
* Histologically or cytologically proven FIGO (International Federation of Gynecology and Obstetrics) stage III to IV epithelial ovarian cancer or peritoneal primary or fallopian tube. A cytological proof is accepted if associated with a ratio of CA125/CEA >25 and a radiological pelvic mass.
* Patient oriented towards a complex medical procedure defined by pelvic surgery preceded or not by antineoplastic treatment (neoadjuvant chemotherapy).
* Therapeutic decision validated in a multidisciplinary consultation meeting
* Life expectancy > 3 months.
* Written informed consent obtained.
* Covered by a Health System where applicable.

Exclusion Criteria:

* Any other progressive malignant tumor interfering with the patient's prognosis.
* Patient whose validated therapeutic management does not include cytoreductive surgery.
* Patient unable to be regularly followed up for any reason (geographic, family, social, psychological).
* Patient unable to understand the questionnaires.
* Patient unable to follow and adhere to test procedures for geographic, social or psychological reasons.
* Patient placed under guardianship or curatorship.
* Patient deprived of liberty.
* Concurrent participation in another interventional drug trial.
* Patient already included in this study

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 292 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2027-06-03 (Estimated); Study Completion 2029-03-03 (Estimated)

PRIMARY OUTCOMES:
Superiority for post-treatment complication grade≥3 | At 30 days post-treatment
  • Superiority for post-treatment complication grade≥3 according the NCI-CTC-v4 (Common Terminology Criteria : CTC) at 30 days
Superiority of HRQOL on the dimensions | At 3 months
  Superiority of HRQOL on the dimensions: Mobility, burden of illness, emotional and physical functioning, fatigue, at 3 months

SECONDARY OUTCOMES:
Post-operative morbidity according Clavien-Dindo classification at 30 and 90 days | At 30 and 90 days
  Clavien Dindo classification consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
  Complications that have the potential for long-lasting disability after patient's discharge (e.g.: paralysis of a voice cord after thyroid surgery) are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a follow-up is required to comprehensively evaluate the outcome and related long-term quality of life.
Therapeutic strategy (treatment plan completion rate) | 2 years
  A complete therapeutic strategy consists of a complete cytoreductive surgery (CC0) 6 courses of chemotherapy at least in total, either in neo-adjuvant or in adjuvant setting, with at least 2 courses after surgery.
Progression free survival | 2 years
  Progression-free survival (PFS) is defined as the time from random assignment to disease progression or death from any cause.
Overall survival | 2 years
  Overall survival is defined as the time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Chu Bordeaux Pellegrin, Bordeaux
  - CH Métropole Savoie, Chambéry
  - Centre Georges François Leclerc, Dijon
  - Hôpital Croix Rousse, Lyon
  - Service de Gériatrie, Centre Hospitalier Lyon Sud, 165 chemin du Grand Revoyet, Pierre-Bénite
  - Centre hospitalier Annecy Genevois, Pringy
  - CHU de St Etienne - Service gynécologie, Saint-Priest-en-Jarez
  - CHU Nord Saint Etienne - Service oncologie médicale, Saint-Priest-en-Jarez
  - Institut Gustave Roussy, Villejuif
  - Médipôle Hôpital Mutualiste, Villeurbanne
  - Villeurbanne Médipole MHP, Villeurbanne